CLINICAL TRIAL: NCT01506635
Title: Effect of Timolol on Refractive Outcomes in Eyes With Myopic Regression After Laser in Situ Keratomileusis: A Randomized Clinical Trial
Brief Title: Effect of Timolol on Refractive Outcomes in Eyes With Myopic Regression After LASIK: a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8902
Record Dates: First submitted 2012-01-04; First posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2009-10

CONDITIONS: Myopic Regression
MeSH Terms: interventions — Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): included patients who received artificial tear twice a day as control group.
  Interventions: Drug: Placebo
- Timolol group (Experimental): included the patients with myopic regression who received timolol 0.5% eye drop twice a day
  Interventions: Drug: Timolol

INTERVENTIONS:
Drug: Timolol
  Arms: Timolol group
Drug: Placebo — artificial tear twice a day
  Arms: Control group

SUMMARY:
In this randomized controlled clinical trial, we compare the effects of timolol versus placebo for treatment of myopic regression after LASIK

ELIGIBILITY:
Inclusion Criteria:

* Patients with myopic regression equal or more than 0.5 D with minimum age of 20 years,
* cylinder ≤ -1.00 D,
* corrected distance visual acuity (CDVA) of at least 20/40 were included.

Exclusion Criteria:

* Patients with a history of previous ocular surgery,
* keratoconus or any ectatic corneal disorder,
* keratoconus suspect by topography,
* preoperative corneal opacity,
* any corneal dystrophies,
* presence of pterygium,
* retinal disorders,
* collagen vascular disorders,
* diabetes mellitus,
* glaucoma,
* cataract,
* pregnancy,
* breast feeding
* systemic corticosteroid therapy were excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Spherical Equivalent | spherical equivalent at month 6
  Effect of timolol use in timolol group will be compared with placebo group at month 6. Moreover, the changes of intragroup spherical equivalent will be assessed in both group 6 months after timolol application.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Shojaei A, Eslani M, Vali Y, Mansouri M, Dadman N, Yaseri M. Effect of timolol on refractive outcomes in eyes with myopic regression after laser in situ keratomileusis: a prospective randomized clinical trial. Am J Ophthalmol. 2012 Nov;154(5):790-798.e1. doi: 10.1016/j.ajo.2012.05.013. Epub 2012 Aug 28. PMID 22935601